CLINICAL TRIAL: NCT03730298
Title: American Ginseng (Panax Quinquefolius) for the Prevention of Moderate-severe Fatigue in Breast Cancer Patients Submitted to Adjuvant Chemotherapy After Surgery. A Study of NICSO (Network Italiano Cure di Supporto in Oncologia).
Brief Title: American Ginseng for the Prevention of Moderate-severe Fatigue in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Network Italiano Cure di Supporto in Oncologia (Other)
Collaborators: Azienda Ospedaliera di Perugia (Other); Associazione Umbra per la lotta Contro il Cancro (Unknown); Avanti Tutta Onlus (Unknown)
Responsible Party: Principal Investigator, Fausto Roila, Medical doctor, Network Italiano Cure di Supporto in Oncologia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICSO-GINSENG
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Cancer Related Fatigue; Breast Cancer Female
Keywords: American Ginseng; Cancer related fatigue; Breast Cancer Female
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- American Ginseng (Experimental): American Ginseng, cpr 700 mg (500 mg of Panax Quinquefolius 5%): 1 cpr twice a day orally for 3 months
  Interventions: Dietary Supplement: American Ginseng
- Placebo (Placebo Comparator): Placebo: 1 cpr twice a day orally for 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: American Ginseng — cpr
  Arms: American Ginseng
Other: Placebo — cpr
  Arms: Placebo

SUMMARY:
Among the symptoms referred by cancer patients, cancer related fatigue (CRF) is one of the most disabling symptom with a relevant impact on the quality of life.

CRF can occur before, during and after anti-cancer treatment. The aim of the present study is to verify the efficacy of American Ginseng in preventing or reducing the intensity of moderate-severe CRF in breast cancer women receiving adjuvant chemotherapy with anthracyclines plus cyclophosphamide after surgery.

DETAILED DESCRIPTION:
Cancer related fatigue (CRF) can occur before, during and after anti-cancer treatment. In fact, up to 40% of patients report fatigue at diagnosis, 80%-90% during chemotherapy and radiotherapy, respectively and 20%-50% in the post-treatment phase.

All cancer patients should be screened for the presence of CRF at the first oncological visit and subsequently during and after the anticancer therapies.

If the patient refers CRF, it could be quantified with one of the validate instruments available; the possible determinants could be identified and corrected if possible, to reduce their impact on patients CR.

The most evaluated pharmacological treatments of CRF include psychostimulants (methylphenidate, modafinil, armodafinil) and dexamethasone. Non-pharmacological treatments include physical exercise, psychological therapies and complementary therapies such as agopuncture, yoga, ginseng.

The aim of the present study is to verify the efficacy of American Ginseng in preventing or reducing the intensity of moderate-severe CRF in a homogeneous population of breast cancer women submitted to adjuvant chemotherapy with anthracyclines plus cyclophosphamide after surgery.

ELIGIBILITY:
Inclusion Criteria:

* submitted for the first time to adjuvant chemotherapy with anthracyclines and cyclophosphamide after surgery for breast cancer;
* not presenting CRF or at least with o al massimo CRF lieve (NRS < 4);
* 18 year old, who have given written informermed consent;
* who accept to use adequate contraceptive methods, if they are of child-bearing potential.

Exclusion Criteria:

* previously submitted to chemotherapy;
* with concomitant not-correctable alterations, present before chemotherapy, possible determinants of fatigue (NRS ≥ 4), such as anemia, not well controlled pain, insomnia, electrolyte imbalance, dehydration, anorexia/cachexia, hepatic, renal or heart failure, adrenocortical failure, neurological deficit, hypothyroidism, not-controlled diabetes mellitus;
* submitted to raitherapy during the 15 days before the randomization;
* presenting moderate-severe fatigue (NRS ≥ 4) at basaline;
* receivind opioids or corticosteroids (except if admimistered at phisiological doses or to prevent emesis on the chemotherapy day);
* with with blood cell count < 3000/mm3, platelets < 70000 mm3, hemoglobin < 8 g/dL;
* unable to understand the procedures of the study or to collaborate with them;
* pregnant or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of cancer related fatigue during chemotherapy. | The NRS will be admistered before randomization (baseline assessment) and before each chemotherapy cycle. In addition, the patients must complete the NRS once a day at home, for 90 days.
  Incidence will be evaluated through the Numeric Rating Scale (NRS). NRS is a linear numeric scale, from 0 = no fatigue to 10 = the worst possible fatigue. A NRS value ≥ 4 indicates the presence of a signficative fatigue (moderate-severe fatigue).
Intensity of cancer related fatigue during chemotherapy. | The NRS will be admistered before randomization (baseline assessment) and before each chemotherapy cycle. In addition, the patients must complete the NRS once a day at home, for 90 days.
  Intensity will be evaluated through the Numeric Rating Scale (NRS). NRS is a linear numeric scale, from 0 = no fatigue to 10 = the worst possible fatigue. A NRS value ≥ 4 indicates the presence of a signficative fatigue (moderate-severe fatigue).moderate-severe fatigue.

SECONDARY OUTCOMES:
Quality of Life (QoL) | These questionnaires will be administered at baseline (before randomization) and immediately before each chemotherapy cycle.
  QoL will be evaluated through validated instruments: the Brief Fatigue Inventory (BFI) and the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-C30), Italian version.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Department, Perugia Hospital, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koornstra RH, Peters M, Donofrio S, van den Borne B, de Jong FA. Management of fatigue in patients with cancer -- a practical overview. Cancer Treat Rev. 2014 Jul;40(6):791-9. doi: 10.1016/j.ctrv.2014.01.004. Epub 2014 Feb 7. PMID 24576643
- [Result] Barton DL, Soori GS, Bauer BA, Sloan JA, Johnson PA, Figueras C, Duane S, Mattar B, Liu H, Atherton PJ, Christensen B, Loprinzi CL. Pilot study of Panax quinquefolius (American ginseng) to improve cancer-related fatigue: a randomized, double-blind, dose-finding evaluation: NCCTG trial N03CA. Support Care Cancer. 2010 Feb;18(2):179-87. doi: 10.1007/s00520-009-0642-2. Epub 2009 May 6. PMID 19415341
- [Result] Barton DL, Liu H, Dakhil SR, Linquist B, Sloan JA, Nichols CR, McGinn TW, Stella PJ, Seeger GR, Sood A, Loprinzi CL. Wisconsin Ginseng (Panax quinquefolius) to improve cancer-related fatigue: a randomized, double-blind trial, N07C2. J Natl Cancer Inst. 2013 Aug 21;105(16):1230-8. doi: 10.1093/jnci/djt181. Epub 2013 Jul 13. PMID 23853057